CLINICAL TRIAL: NCT03268967
Title: Optimized Admission to the Intensive Care Unit by Using Crisis Resource Management (CRM)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hillerod Hospital, Denmark (Other)
Collaborators: Holbaek Sygehus (Other)
Responsible Party: Principal Investigator, Janet Froulund Jensen, PHD, Principal Investigator, Hillerod Hospital, Denmark
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: 113581; 113581 (Other Grant/Funding Number: Trygfonden)
Record Dates: First submitted 2017-08-28; First posted 2017-08-31 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Critical Illness
Keywords: intensive care; crisis resource management; simulation training; before and after study
MeSH Terms: conditions — Critical Illness | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Before and after interventional study
Who Masked: Outcomes Assessor
Masking Description: Data analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured Admission procedure (Active Comparator): After implementation of a structured admission procedure to all ICU patients inspired by principles of Crisis Resource Management, Closed loop communication, action cards, and staff simulation training
  Interventions: Behavioral: Structured admission procedure
- Standard Care (No Intervention): Randomly admission procedure to all ICU patients based on the clinicians' evaluation prior implementation of the intervention.

INTERVENTIONS:
Behavioral: Structured admission procedure — A structured ICU admission was inspired by principles of Crisis Resource Management and simulation training of ICU staff members. The Principles of Crisis Resource Management consisted of a treatment manual, a learning video, clear precise communication tool based on Identification-Situation-Background-Analysis-Recommendations (ISBAR) and Closed loop, actions cards, and ABCDE-evaluation of the patient including debriefing, and training in the simulation environment.
  Other Names: Standard Care
  Arms: Structured Admission procedure

SUMMARY:
Admission to the intensive care unit (ICU) is vital for surviving critical illness. An admission to ICU without having a consistent structure, structured review of the patient and a solid team organization lead to unclear communication and responsibility. Factors that correlate with patient acceptance and safety, morbidity and mortality. The hypothesize was that a structured admission can improve patients safety, reduce delays in treatment, reduce ICU length of stay, and improve mortality rate. The overall objective was to optimize patient safety, and effectively use available resources to reduce admission time, delays in treatment and procedures and mortality by using both quantitative and qualitative methods.

DETAILED DESCRIPTION:
The quantitative before-data is a one-year observational period prior to the intervention measured by different perspectives; patients and staff outcomes.

After the intervention, was qualititive data collected from participants, who received simulation training.

The quantitative after-data is a one-year observational period post-intervention with same outcomes as before starting the intervention.

Data is already collected registry data from hospital quality assurance board. Data will be compared before and after with assessor blinded analysis. Missing data will not be replaced but reported as missing.

The investigators will try to compare the results with data from an approximately comparative ICU in Denmark due to the implementation of a new patient management system called the Health Portal.

The statistical analysis plan is based on descriptive and comparative analyses of the group before and after the trial. The quantitative results are explained in in-depths description from participants.

ELIGIBILITY:
Inclusion Criteria:

* ICU admissions

Exclusion Criteria:

* None
* Drop-out are deaths

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2014-04-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
ICU length of stay (LOS) | through study completion, an average of 1 year
  Days admitted at the ICU using registre data

SECONDARY OUTCOMES:
Hospital length of stay (LOS) | At Hospital discharge within one-year before and after the intervention implementation
  Days admitted to the hospital using registre data
Line Sepsis | through study completion, an average of 1 year
  Treatment package of number of the line sepsis after ICU admission covering the number of patients with line sepsis using registre data on Lactat <1 hour, bacteria samples ≤1 hour taken, time between diagnosis of sepsis and taken bacteria samples, time between diagnosis and given antibiotics measured by registre data
Ventilated associated pneumonia (VAP) | through study completion, an average of 1 year
  Number of VAP measured by registre data
Re-intubations | through study completion, an average of 1 year
  Number of re-intubations measured by registre data
30-days Mortality | 30 days through study completion, an average of 1 year
  30-days mortality rates after ICU discharge measured by registre data
90-days Mortality | 90 days through study completion, an average of 1 year
  90-days mortality rates after ICU discharge measured by registre data
Staff turn-over | through study completion, an average of 1 year
  Staff turn-over before and after the intervention measured by registre data
Sick Leave | through study completion, an average of 1 year
  Sick leave amongst staff members measured by registre data

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaestesiology, Holbæk, Denmark

IPD SHARING:
Plan to Share IPD: Undecided